CLINICAL TRIAL: NCT07060326
Title: Digital Literacy in Caregivers of Pediatric Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Brittany Willer (Other)
Responsible Party: Sponsor-Investigator, Brittany Willer, Pediatric Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00004951
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Digital Literacy; Pediatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents / Caregivers: Parents / caregivers of pediatric patients presenting for surgery.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — REDCap Survey

SUMMARY:
The purpose of this study is to describe the digital literacy of caregivers of pediatric surgical patients. The investigators hypothesize that caregivers of minority race, language of care other than English, and low neighborhood opportunity will have lower prevalence of digital literacy.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children <18 presenting for surgery at NCH. Primary language must be English, Spanish, Arabi, Nepali, or Somali.

Exclusion Criteria:

* Patients who are 18 years of age or older. Wards of the state. Patients who are missing address information.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Caregivers of children <18 presenting for surgery at NCH.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
EDLQ digital literacy scores | From enrollment to end of perioperative time.

SECONDARY OUTCOMES:
eHEALS Health Literacy scores | From enrollment to end of perioperative time.
  eHEALS Health Literacy scores across three domains: information and communication, content creation and management, safety and security.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No